CLINICAL TRIAL: NCT02857413
Title: Assessment of Frequency of Xerostomia and Their Care Management in Upper Aerodigestive Tract Cancer Patients After the End of Radiotherapy
Brief Title: Frequency of Xerostomia and Their Management in Upper Aerodigestive Tract Cancer Patients After the End of Radiotherapy
Acronym: XEROSTOMIA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2015/281
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Head and Neck Neoplasms
Keywords: Xerostomia; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is the evaluation of the frequency of xerostomia and their management after radiotherapy in head and neck cancer.

The quality of life of these patients is also analysed with European Organization for Research and Treatment of Cancer Quality of life Questionnaire H&N35 (EORTC QLQ H&N35).

ELIGIBILITY:
Inclusion Criteria:

* patient with head and neck cancer after radiotherapy treatment

Exclusion Criteria:

* patient already treated for xerostomia for other reason : Sjögren's syndrome, medication, diabetes,...

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with head and neck cancer after radiotherapy treatment
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Frequency of xerostomia and their management after radiotherapy in head and neck cancer | at enrollment
  patients describe the severity of their xerostomia and their management in a standardized questionnaire

SECONDARY OUTCOMES:
quality of life af patients after radiotherapy in head and neck cancer | at enrollment
  patients describe their quality of life in a standardized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Euvrard, MD, Principal Investigator — CHU Besançon
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No